CLINICAL TRIAL: NCT06581276
Title: Increasing Access to Evidence-based Treatment for Chronic Pain and Opioid Use Disorder: Adapting Acceptance and Commitment Therapy for Opioid Treatment Programs
Acronym: OTP-ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-14272
Record Dates: First submitted 2024-08-27; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Opioid Use; Opioid Use Disorder; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OTP Intervention (Other): Evidence-based behavioral pain treatment integrated into OTP model of care
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — Acceptance and Commitment Therapy (ACT) is an evidence-based behavioral pain treatment intervention for Chronic Pain, anxiety and depression, and substance use disorders, being studied as a group-based therapy delivered by substance use counselors in an opioid treatment program.

SUMMARY:
The overarching goal of this study was to provide patient-centered treatment for chronic pain in opioid treatment programs (OTPs). Chronic pain (CP) is highly prevalent among people with opioid use disorder (OUD) who attend OTPs, with 64% of OTP patients experiencing CP and 37% reporting severe CP. OTP patients are required to attend programs frequently for medication administration, which makes the OTP an ideal location to deliver pain treatment; however, in a large national survey of people entering OUD treatment, only one-third of patients had CP treated in their program. People with OUD attending OTPs are highly marginalized and may lack access to multimodal pain management and mental health services. Integrating evidence-based treatments for CP and its associated comorbidities (such as anxiety and depression) into OTPs could have broad impact.

DETAILED DESCRIPTION:
Training OTP counselors to deliver evidence-based pain interventions may be the ideal way to integrate pain and OUD treatment. There is a strong tradition of OTP counselors providing individual and group counseling, but it is typically focused on substance use recovery. Acceptance and Commitment Therapy (ACT), an evidence-based intervention for CP, anxiety and depression, and substance use disorders, is being studied in the IMPOWR-ME center as a group-based therapy combined with outpatient buprenorphine treatment for delivery in the primary care setting. Successful delivery of ACT in OTPs would require modifying its content and format to meet the needs of the OTP setting and patients. IMPOWR-ME's ACT is a 12-session, psychologist-led intervention. ACT has been effectively delivered by lay-person facilitators and many OTP counselors are accustomed to on-the-job training. However one modifiable barrier is that OTP counselors primarily work from an abstinence-based model, which is in conflict with ACT principles (i.e. patients identifying their own values and goals). Although OTPs have a longstanding commitment to running groups, group ACT, with its structured and sequential content, may run counter to OTP norms of open attendance and unstructured discussion. Notable OTP attendance barriers such as transportation and competing priorities may also hinder completion of 12-session protocols like that of the IMPOWR-ME trial.

To address these challenges, the investigator team: 1) Trained OTP counselors to deliver ACT and provided ongoing supervision; 2) Increased OTP counselors' familiarity and technical skill in harm reduction counseling strategies (patient-identified goal setting and monitoring) to complement ACT principles; 3) Adapted ACT's format and content to be culturally aligned with OTP patients (including language, concepts and metaphors) and responsive to the needs and preferences of OTP patients for group therapy (number of sessions, use of sequential content). Perspectives of OTP patients and staff were incorporated. The 12-month pilot study consisted of the following 3 Aims:

Aim 1: Adapted the IMPOWR-ME high-intensity ACT intervention to meet the needs of an OTP. Guided by the Center for Disease Control and Prevention (CDC) framework for adapting evidence-based interventions and Bernal's ecological validity model, the investigator team developed a modified ACT protocol in collaboration with the IMPOWR-ME ACT team, content experts, and OTP stakeholders. Two stakeholder studios (1 with OTP staff, 1 with OTP patients) provided input on how to adapt ACT for optimal feasibility and acceptability for OTP patients. With the IMPOWR-ME ACT team and content experts, the investigator team systematically modified ACT structure and content to address stakeholder studio recommendations. Then, 4 OTP counselors interested in serving as ACT group leaders were recruited and trained in the adapted ACT protocol.

Aim 2: Examined feasibility and acceptability of adapted ACT in an OTP and study OTP counselor fidelity to the intervention: 15 patients were recruited and enrolled to pilot the adapted ACT intervention during one of two, 12-session groups. To assess feasibility, the study team used qualitative data from in-depth interviews with OTP ACT group leaders on time, skills, and other resources required to deliver the intervention. To assess the acceptability of the intervention, the study team conducted questionnaires and in-depth interviews with patients to examine their experiences with and attitudes toward the intervention and suggestions for modifications (N=15). The investigator team examined the acceptability of the intervention to the ACT group leaders during in-depth qualitative interviews at the end of the study (N=3). ACT group leader fidelity to key principles of ACT facilitation and harm reduction principles was rated for 6 video recorded group sessions.

Aim 3, the basis of this registration, was conducted to examine changes in patient non-prescription opioid use, overdose risk behavior, anxiety, depression, pain interference, pain catastrophizing and pain acceptance pre and post-intervention. The study team administered baseline and follow-up questionnaires upon completion of the ACT intervention to assess changes in clinical outcomes. Completion of these aims provides a manual for group-based ACT for CP and OUD in OTPs and data on the feasibility and acceptability of providing ACT in OTPs. This data is going to be used to apply for a National Institute on Drug Abuse (NIDA) R34 grant to plan a Randomized Control Trial (RCT) studying the effectiveness of ACT for CP and OUD outcomes among OTP participants.

ELIGIBILITY:
Inclusion Criteria:

* Opioid Treatment Program (OTP) patients;
* Patient self-report of at least moderate Chronic Pain of any duration;
* Willingness to participate in video-recorded ACT group sessions to be viewed by the study team
* Fluent in English

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Change in Non-Prescription Opioid Use | Pre-Intervention and Post-Intervention, approximately 12 weeks
  Change in Non-Prescription Opioid Use from Pre-intervention to Post-intervention will be assessed by administration of the Addiction Severity Index (ASI) to OTP participants at enrollment and upon completion of the ACT session. The ASI is a structured clinical interview consisting of 7 statements asking patients about opioid use over the last 30 days and their lifetime. For this study, each item is scored such that if the patient answers "Yes" they may score 1; if they answer "No", they may score 0. For some items, the scoring may be reversed. A composite score is used to assign a severity rating. Basic descriptive statistics will be used to summarize group results. Negative group mean scores are associated with a lowered need for opioid treatment following intervention and positive group mean scores are associated with an increased need for opioid treatment following intervention.
Change in Overdose Risk Behavior | Pre-Intervention and Post-Intervention, approximately 12 weeks
  Change in Overdose Risk Behavior from Pre-intervention to Post-intervention will be assessed using a modification of the Opioid Risk Behavior Scale (ORBS2). This 26-item instrument tailored to each patient's use of substances selected from a screening question containing opioid and opioid-contraindicated categories. Concurrent use of opioids and other contraindicated substances are generated based on the specific drugs selected from the list and progress from combinations as indicated on the form. Pictures of the substances are included to aid participants in identifying the polysubstance combinations. Patients are asked to identify the number of days within the past 30 days they engaged in each activity. Scores are summarized for an overall possible score of 0-780. Basic descriptive statistics will be used to summarize group results. Negative group mean scores are associated with decreased overdose risk behavior following intervention and positive group mean scores are associated
Change in Anxiety | Pre-Intervention and Post-Intervention, approximately 12 weeks
  Change in Anxiety from Pre-intervention to Post-intervention will be assessed using the General Anxiety Disorder (GAD-7) scale. The GAD-7 is a 7-item self-report anxiety scale consisting of 7 statements asking patients to rate how often they have been bothered by the problems identified within each statement over the prior 2 weeks. Each item is scored on a 4-point scale ranging from 0 ("Not at all sure") to 3 ("Nearly every day") yielding an overall possible score of 0-21. Basic descriptive statistics will be used to summarize group results. Negative group mean scores are associated with decreased severity of anxiety following intervention and positive group mean scores are associated with increased severity of anxiety following intervention.
Change in Depression | Pre-Intervention and Post-Intervention, approximately 12 weeks
  Change in Depression from Pre-intervention to Post-intervention will be assessed using the 9-item Patient Health Questionnaire (PHQ-9). The PHQ-9 is a 9-item self-report depression severity scale consisting of 9 statements asking patients to rate how often they have been bothered by the problems within each statement over the prior 2 weeks. Each item is scored on a 4-point scale ranging from 0 ("Not at all") to 3 ("Nearly every day") yielding an overall possible score of 0-27. Basic descriptive statistics will be used to summarize group results. Negative group mean scores are associated with lower depression severity following intervention and positive group mean scores are associated with greater depression severity following intervention.
  The PHQ-9 also includes a single screening question about suicide risk however this question is not part of the Outcome Measures for this study.
Change in Pain Intensity and Interference - PEG | Pre-Intervention and Post-Intervention, approximately 12 weeks
  Change in Pain Interference from Pre-intervention to Post-intervention will be assessed using the Pain, Enjoyment, General Activity (PEG) scale. The PEG scale is a 3-item, patient-reported pain scale used to assess and monitor chronic pain intensity and interference. The scale is based on the Brief Pain Inventory and consists of three numerical scales (Pain on average over the past week'; 'Enjoyment of Life'; and 'Pain Interference of general activities') each ranging from 0 ("No Pain" or "Does not interfere") to 10 ("Pain as bad as you can imagine" or "Completely interferes"). Basic descriptive statistics will be used to summarize group results from the three scales for an overall possible range of 0-30. Negative group mean scores are associated with a reduction in pain intensity and interference following intervention and positive group mean scores are associated with an increase in pain intensity and interference following intervention.
Change in Pain Interference - Patient-Reported Outcomes Measurement Information System (PROMIS) | Pre-Intervention and Post-Intervention, approximately 12 weeks
  Change in Pain Interference from Pre-intervention to Post-intervention will also be assessed using the PROMIS Pain Interference - Short Form 8a. This 8-item scale which measures the self-reported consequences of pain on relevant aspects of a person's life asks patients to respond how often pain interfered with universal activities over the prior 7 day period on a 5-point scale ranging from 1 ("Not at all") to 5 ("Very much") yielding an overall possible score of 8-40. Basic descriptive statistics will be used to summarize group results. Negative group mean scores are associated with a reduction in pain interference during the conduct of universal activities following intervention and positive group mean scores are associated with an increase in pain interference during the conduct of universal activities following intervention.
Change in Pain Catastrophizing | Pre-Intervention and Post-Intervention, approximately 12 weeks
  Change in Pain Catastrophizing from Pre-intervention to Post-intervention will be assessed using the Pain Catastrophizing Scale (PCS). The PCS is a 13-item self-report questionnaire that asks patients to rate how often they experience certain thoughts and feelings when in pain and span the categories of rumination, magnification, and helplessness. Each item is scored on a 5-point scale ranging from 0 ("Not at all") to 4 ("All the time") yielding an overall possible score of 0-52. Basic descriptive statistics will be used to summarize group results. Negative group mean scores are associated with a reduction in pain catastrophizing following intervention and positive group mean scores are associated with an increase in pain catastrophizing following intervention.
Change in Pain Acceptance | Pre-Intervention and Post-Intervention, approximately 12 weeks
  Change in Pain Acceptance from Pre-intervention to Post-intervention will be assessed using the Chronic Pain Acceptance Questionnaire - Revised (CPAQ-R). The CPAQ-R consists 20 of statements asking the patient to rate the truth of each statement on a 7-point Likert scale ranging from 0 ("Never true") to 6 ("Always true") for an overall possible range of 0-120. Basic descriptive statistics will be used to summarize group results. Positive group mean scores are associated with improvement in pain acceptance following intervention and negative group scores are associated with a decrease in pain acceptance following intervention.
Satisfaction with Treatment | Pre-Intervention and Post-Intervention, approximately 12 weeks
  Patient satisfaction with treatment was assessed using the Patients' Global Impression of Change (PGIC) Scale. The PGIC consists of a single question asking the patient how they would describe the change (if any) in Activity, Limitations, Symptoms, Emotions, and overall Quality of Life (QoL) related to their condition following the intervention. A response is provided based on a 7-point Likert scale ranging from 1 ("No Change") to 7 ("A great deal better") for an overall possible range of 1-7. Higher scores are associated with overall improvement in condition. Basic descriptive statistics will be used to summarize group results.
Problematic Substance Use | Pre-Intervention and Post-Intervention, approximately 12 weeks
  Change in problematic substance use was assessed using the Short Inventory of Problems Alcohol and Drugs (SID-AD), a fifteen-item instrument asking patients to rate how often they have experienced a range of problems related to alcohol and/or drug use during the past 30 days. Each item is scored on a 4-point scale ranging from 0 ("Never") to 3 ("Daily or almost daily"), yielding an overall possible score of 0-45. Basic descriptive statistics will be used to summarize group results. Negative group mean scores are associated with reductions in problematic substance use following intervention.
Psychological flexibility | Pre-Intervention and Post-Intervention, approximately 12 weeks
  Change in psychological flexibility was assessed using the Multidimensional Psychological Flexibility Inventory (MPFI-12). The MPFI-12 is a 12-item scale with six items assessing psychological flexibility, and six items assessing psychological inflexibility. Patients are asked about responses to thoughts, feelings, and actions aligned with their values on a 6-point scale ranging from 1 ("Never true") to 6 ("Always true"), yielding an overall possible score of 6-36 for flexibility and 6-36 for inflexibility. Basic descriptive statistics will be used to summarize group results. Positive group mean scores for flexibility and negative group mean scores for inflexibility are associated with improvement following intervention.
Committed Action | Pre-Intervention and Post-Intervention, approximately 12 weeks
  Change in committed action was assessed using the committed Action Questionnaire (CAQ). The CAQ is an 18-item measure asking patients to indicate agreement with statements about how they take goal-directed actions ranging from 0 ("never true") to 6 ("always true"), yielding a score of 0-108. Basic descriptive statistics will be used to summarize group results. Positive group mean scores for committed action are associated with improvement following the intervention.
Acceptance and Action Related to Substance Use | Pre-Intervention and Post-Intervention, approximately 12 weeks
  Change in acceptance and actions related to substance use were assessed using the Acceptance and Action Questionnaire for Substance Abuse (AAQSA). The AAQSA is an 18-item measure asking patients to indicate responses to thoughts and feelings about their substance use from 1 ("never true") to 7 ("always true"), yielding an overall possible score of 18- 126. Basic descriptive statistics will be used to summarize group results. Positive group mean scores for acceptance and action are associated with improvement following the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Jakubowski, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center Division of General Internal Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hser YI, Mooney LJ, Saxon AJ, Miotto K, Bell DS, Huang D. Chronic pain among patients with opioid use disorder: Results from electronic health records data. J Subst Abuse Treat. 2017 Jun;77:26-30. doi: 10.1016/j.jsat.2017.03.006. Epub 2017 Mar 9. PMID 28476267
- [Background] Rosenblum A, Joseph H, Fong C, Kipnis S, Cleland C, Portenoy RK. Prevalence and characteristics of chronic pain among chemically dependent patients in methadone maintenance and residential treatment facilities. JAMA. 2003 May 14;289(18):2370-8. doi: 10.1001/jama.289.18.2370. PMID 12746360
- [Background] Ellis MS, Kasper Z, Cicero T. Assessment of Chronic Pain Management in the Treatment of Opioid Use Disorder: Gaps in Care and Implications for Treatment Outcomes. J Pain. 2021 Apr;22(4):432-439. doi: 10.1016/j.jpain.2020.10.005. Epub 2020 Nov 14. PMID 33197581
- [Background] Han BH, Doran KM, Krawczyk N. National trends in substance use treatment admissions for opioid use disorder among adults experiencing homelessness. J Subst Abuse Treat. 2022 Jan;132:108504. doi: 10.1016/j.jsat.2021.108504. Epub 2021 May 29. PMID 34102461
- [Background] Lee C, Crawford C, Swann S; Active Self-Care Therapies for Pain (PACT) Working Group. Multimodal, integrative therapies for the self-management of chronic pain symptoms. Pain Med. 2014 Apr;15 Suppl 1:S76-85. doi: 10.1111/pme.12408. PMID 24734863
- [Background] Hughes LS, Clark J, Colclough JA, Dale E, McMillan D. Acceptance and Commitment Therapy (ACT) for Chronic Pain: A Systematic Review and Meta-Analyses. Clin J Pain. 2017 Jun;33(6):552-568. doi: 10.1097/AJP.0000000000000425. PMID 27479642
- [Background] Coto-Lesmes R, Fernandez-Rodriguez C, Gonzalez-Fernandez S. Acceptance and Commitment Therapy in group format for anxiety and depression. A systematic review. J Affect Disord. 2020 Feb 15;263:107-120. doi: 10.1016/j.jad.2019.11.154. Epub 2019 Dec 2. PMID 31818766
- [Background] Lee EB, An W, Levin ME, Twohig MP. An initial meta-analysis of Acceptance and Commitment Therapy for treating substance use disorders. Drug Alcohol Depend. 2015 Oct 1;155:1-7. doi: 10.1016/j.drugalcdep.2015.08.004. Epub 2015 Aug 13. PMID 26298552
- [Background] Purgato M, Carswell K, Tedeschi F, Acarturk C, Anttila M, Au T, Bajbouj M, Baumgartner J, Biondi M, Churchill R, Cuijpers P, Koesters M, Gastaldon C, Ilkkursun Z, Lantta T, Nose M, Ostuzzi G, Papola D, Popa M, Roselli V, Sijbrandij M, Tarsitani L, Turrini G, Valimaki M, Walker L, Wancata J, Zanini E, White R, van Ommeren M, Barbui C. Effectiveness of Self-Help Plus in Preventing Mental Disorders in Refugees and Asylum Seekers in Western Europe: A Multinational Randomized Controlled Trial. Psychother Psychosom. 2021;90(6):403-414. doi: 10.1159/000517504. Epub 2021 Jul 20. PMID 34350902
- [Background] Acarturk C, Uygun E, Ilkkursun Z, Carswell K, Tedeschi F, Batu M, Eskici S, Kurt G, Anttila M, Au T, Baumgartner J, Churchill R, Cuijpers P, Becker T, Koesters M, Lantta T, Nose M, Ostuzzi G, Popa M, Purgato M, Sijbrandij M, Turrini G, Valimaki M, Walker L, Wancata J, Zanini E, White RG, van Ommeren M, Barbui C. Effectiveness of a WHO self-help psychological intervention for preventing mental disorders among Syrian refugees in Turkey: a randomized controlled trial. World Psychiatry. 2022 Feb;21(1):88-95. doi: 10.1002/wps.20939. PMID 35015365
- [Background] Mercer, D. E., D, P. & Woody, G. E. Individual Drug Counseling. in Therapy Manuals for Drug Addiction Series 1-77 (U.S. Department of Health and Human Services, NIH, NIDA, 1999)
- [Background] McKleroy VS, Galbraith JS, Cummings B, Jones P, Harshbarger C, Collins C, Gelaude D, Carey JW; ADAPT Team. Adapting evidence-based behavioral interventions for new settings and target populations. AIDS Educ Prev. 2006 Aug;18(4 Suppl A):59-73. doi: 10.1521/aeap.2006.18.supp.59. PMID 16987089
- [Background] Bernal G, Bonilla J, Bellido C. Ecological validity and cultural sensitivity for outcome research: issues for the cultural adaptation and development of psychosocial treatments with Hispanics. J Abnorm Child Psychol. 1995 Feb;23(1):67-82. doi: 10.1007/BF01447045. PMID 7759675
- [Background] Alderks CE. Trends in the Use of Methadone, Buprenorphine, and Extended-Release Naltrexone at Substance Abuse Treatment Facilities: 2003-2015 (Update). 2017 Aug 22. In: The CBHSQ Report. Rockville (MD): Substance Abuse and Mental Health Services Administration (US); 2013-. Available from http://www.ncbi.nlm.nih.gov/books/NBK469748/ PMID 29200242
- [Background] Heimer R, Zhan W, Grau LE. Prevalence and experience of chronic pain in suburban drug injectors. Drug Alcohol Depend. 2015 Jun 1;151:92-100. doi: 10.1016/j.drugalcdep.2015.03.007. Epub 2015 Mar 19. PMID 25841984
- [Background] Kelly SM, Schwartz RP, O'grady KE, Gandhi D, Jaffe JH. Impact of methadone with versus without drug abuse counseling on HIV risk: 4- and 12-month findings from a clinical trial. J Addict Med. 2012 Jun;6(2):145-52. doi: 10.1097/ADM.0b013e31823ae556. PMID 22134175
- [Background] Schwartz RP, Kelly SM, O'Grady KE, Gandhi D, Jaffe JH. Interim methadone treatment compared to standard methadone treatment: 4-month findings. J Subst Abuse Treat. 2011 Jul;41(1):21-9. doi: 10.1016/j.jsat.2011.01.008. Epub 2011 Feb 24. PMID 21353445
- [Background] Daley, D. C., Mercer, D. & Carpenter, G. Drug counseling for cocaine addiction: The Collaborative Cocaine Treatment Study Model. in Trastornos Adictivos (U.S. Department of Health and Human Services, NIH, NIDA, 2002). doi:10.1016/s1575-0973(03)70109-3
- [Background] Collins, S. Harm Reduction Training for Substance Use: Meeting people where they're at. (2017). Available at: https://aims.uw.edu/ictp/Harm_Reduction_Training_Susan_Collins_PhD_08-17-2017.pdf.
- [Background] Collins SE, Duncan MH, Saxon AJ, Taylor EM, Mayberry N, Merrill JO, Hoffmann GE, Clifasefi SL, Ries RK. Combining behavioral harm-reduction treatment and extended-release naltrexone for people experiencing homelessness and alcohol use disorder in the USA: a randomised clinical trial. Lancet Psychiatry. 2021 Apr;8(4):287-300. doi: 10.1016/S2215-0366(20)30489-2. Epub 2021 Mar 10. PMID 33713622
- [Background] Collins SE, Clifasefi SL, Nelson LA, Stanton J, Goldstein SC, Taylor EM, Hoffmann G, King VL, Hatsukami AS, Cunningham ZL, Taylor E, Mayberry N, Malone DK, Jackson TR. Randomized controlled trial of harm reduction treatment for alcohol (HaRT-A) for people experiencing homelessness and alcohol use disorder. Int J Drug Policy. 2019 May;67:24-33. doi: 10.1016/j.drugpo.2019.01.002. Epub 2019 Mar 6. PMID 30851620
- [Background] Mitchell SG, Monico LB, Lertch E, Kelly SM, Gryczynski J, Jaffe JH, O'Grady KE, Schwartz RP. Counseling Staff's Views of Patient-Centered Methadone Treatment: Changing Program Rules and Staff Roles. J Behav Health Serv Res. 2018 Jul;45(3):506-515. doi: 10.1007/s11414-018-9603-1. PMID 29536342
- [Background] New York City Department of Health and Mental Hygiene. Epi Data Brief: Unintentional Drug Poisoning (Overdose) Deaths in New York City in 2018. (2019).
- [Background] Torres Blasco N, Costas Muniz R, Zamore C, Porter L, Claros M, Bernal G, Shen MJ, Breitbart W, Castro EM. Cultural adaptation of meaning-centered psychotherapy for latino families: a protocol. BMJ Open. 2022 Apr 4;12(4):e045487. doi: 10.1136/bmjopen-2020-045487. PMID 35379609
- [Background] Mabunda D, Oliveira D, Sidat M, Cavalcanti MT, Cumbe V, Mandlate F, Wainberg M, Cournos F, de Jesus Mari J. Cultural adaptation of psychological interventions for people with mental disorders delivered by lay health workers in Africa: scoping review and expert consultation. Int J Ment Health Syst. 2022 Feb 15;16(1):14. doi: 10.1186/s13033-022-00526-x. PMID 35168650
- [Background] Venner KL, Hernandez-Vallant A, Hirchak KA, Herron JL. A scoping review of cultural adaptations of substance use disorder treatments across Latinx communities: Guidance for future research and practice. J Subst Abuse Treat. 2022 Jun;137:108716. doi: 10.1016/j.jsat.2021.108716. Epub 2022 Jan 11. PMID 35148923
- [Background] Stallings SC, Boyer AP, Joosten YA, Novak LL, Richmond A, Vaughn YC, Wilkins CH. A taxonomy of impacts on clinical and translational research from community stakeholder engagement. Health Expect. 2019 Aug;22(4):731-742. doi: 10.1111/hex.12937. Epub 2019 Jul 18. PMID 31321849
- [Background] Joosten YA, Israel TL, Williams NA, Boone LR, Schlundt DG, Mouton CP, Dittus RS, Bernard GR, Wilkins CH. Community Engagement Studios: A Structured Approach to Obtaining Meaningful Input From Stakeholders to Inform Research. Acad Med. 2015 Dec;90(12):1646-50. doi: 10.1097/ACM.0000000000000794. PMID 26107879
- [Background] O'Neill, L., Latchford, G., McCracken, L. M. & Graham, C. D. The development of the Acceptance and Commitment Therapy Fidelity Measure (ACT-FM): A delphi study and field test. J. Context. Behav. Sci. 14, 111-118 (2019).
- [Background] Collins, S. E. & Cilasefi, S. L. Harm Reduction Approaches | Advances in Psychotherapy: Evidence-Based Practice, Volume 52. (Hogrefe Publishing, 2023).
- [Background] Kelly PJ, Kyngdon F, Ingram I, Deane FP, Baker AL, Osborne BA. The Client Satisfaction Questionnaire-8: Psychometric properties in a cross-sectional survey of people attending residential substance abuse treatment. Drug Alcohol Rev. 2018 Jan;37(1):79-86. doi: 10.1111/dar.12522. Epub 2017 May 7. PMID 28480521
- [Background] Nowell, L. S., Norris, J. M., White, D. E. & Moules, N. J. Thematic Analysis: Striving to Meet the Trustworthiness Criteria. Int. J. Qual. Methods 16, 1-13 (2017).
- [Background] McLellan AT, Luborsky L, Woody GE, O'Brien CP. An improved diagnostic evaluation instrument for substance abuse patients. The Addiction Severity Index. J Nerv Ment Dis. 1980 Jan;168(1):26-33. doi: 10.1097/00005053-198001000-00006. PMID 7351540
- [Background] Elliott L, Crasta D, Khan M, Roth A, Green T, Kolodny A, Bennett AS. Validation of the Opioid Overdose Risk Behavior Scale, version 2 (ORBS-2). Drug Alcohol Depend. 2021 Jun 1;223:108721. doi: 10.1016/j.drugalcdep.2021.108721. Epub 2021 Apr 20. PMID 33895681
- [Background] Weiss L, Egan JE, Botsko M, Netherland J, Fiellin DA, Finkelstein R. The BHIVES collaborative: organization and evaluation of a multisite demonstration of integrated buprenorphine/naloxone and HIV treatment. J Acquir Immune Defic Syndr. 2011 Mar 1;56 Suppl 1:S7-13. doi: 10.1097/QAI.0b013e3182097426. PMID 21317598